CLINICAL TRIAL: NCT02729090
Title: Effects of Combined Force Training Aerobic Versus Aerobic in the Functional Capacity, Central Artery and Rigidity Ankle Brachial Index in Patients With Peripheral Artery Disease
Brief Title: Effects of Exercise in the Functional Capacity, Central Artery and Rigidity Ankle Brachial Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0381
Record Dates: First submitted 2016-02-18; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease, exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device: treadmill (Experimental): Aerobic training on a treadmill continuously with speed and wave periodization. Frequency twice per week ( 2x ) for twelve weeks
  Interventions: Other: Device: treadmill
- Device: treadmill Train_Comb_aerobic (Active Comparator): strength training with free weights, followed by active recovery on a treadmill with fixed intervals of 60 to 120 seconds between each workforce of series.
  Interventions: Other: Device: treadmill Train_Comb_aerobic

INTERVENTIONS:
Other: Device: treadmill — Aerobic training on a treadmill continuously with speed and wave periodization. Frequency twice per week ( 2x ) for twelve weeks. Device: treadmill.
  Arms: Device: treadmill
Other: Device: treadmill Train_Comb_aerobic — Device: treadmill Train_Comb_aerobic. strength training with free weights, followed by active recovery on a treadmill with fixed intervals of 60 to 120 seconds between each workforce of series. Device: treadmill Train_Comb_aerobic
  Arms: Device: treadmill Train_Comb_aerobic

SUMMARY:
The Peripheral Arterial Disease prevalence is around 3-10 % of the world population. Exercise plays an important role in treating these patients.

DETAILED DESCRIPTION:
Objective: To investigate the effects of training Combined Aerobic - Strength versus aerobic functional capacity, ankle brachial index (ABI ) and central arterial stiffness in patients with peripheral arterial disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DAP and CI .
* Stage I or II of Fontaine .
* intermittent claudication symptoms for at least 3 months with ankle brachial index (ABI ) at rest ≤ 0.90 in 1 or 2 legs.

Exclusion Criteria:

* Ischemia criticism in one of the lower limbs.
* moderate or severe ulcers on one of the lower limbs.Orthopedic issues that prevent pratical of the exercises or conducting evaluations .
* Participation in other studies with rehabilitation.
* decompensated hypertension .
* decompensated diabetes .
* Cardiovascular events less than three months .
* severe lung disease .

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary test - 6 minute walk test | 48 months
  evaluation of functional capacity

SECONDARY OUTCOMES:
Pulse wave velocity | 48 months
One maximum repetition test | 48 months
ankle brachial index | 48 months
Edinburgh Claudication Questionnaire | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. Dos Santos, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital De Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rehring TF, Sandhoff BG, Stolcpart RS, Merenich JA, Hollis HW Jr. Atherosclerotic risk factor control in patients with peripheral arterial disease. J Vasc Surg. 2005 May;41(5):816-22. doi: 10.1016/j.jvs.2005.01.047. PMID 15886666
- [Background] Rabkin SW, Chan SH, Sweeney C. Ankle-brachial index as an indicator of arterial stiffness in patients without peripheral artery disease. Angiology. 2012 Feb;63(2):150-4. doi: 10.1177/0003319711410307. Epub 2011 Jun 15. PMID 21676966
- [Background] Laurent S, Boutouyrie P, Asmar R, Gautier I, Laloux B, Guize L, Ducimetiere P, Benetos A. Aortic stiffness is an independent predictor of all-cause and cardiovascular mortality in hypertensive patients. Hypertension. 2001 May;37(5):1236-41. doi: 10.1161/01.hyp.37.5.1236. PMID 11358934
- [Background] McDermott MM, Ades P, Guralnik JM, Dyer A, Ferrucci L, Liu K, Nelson M, Lloyd-Jones D, Van Horn L, Garside D, Kibbe M, Domanchuk K, Stein JH, Liao Y, Tao H, Green D, Pearce WH, Schneider JR, McPherson D, Laing ST, McCarthy WJ, Shroff A, Criqui MH. Treadmill exercise and resistance training in patients with peripheral arterial disease with and without intermittent claudication: a randomized controlled trial. JAMA. 2009 Jan 14;301(2):165-74. doi: 10.1001/jama.2008.962. PMID 19141764
- [Background] Wang J, Zhou S, Bronks R, Graham J, Myers S. Effects of supervised treadmill walking training on calf muscle capillarization in patients with intermittent claudication. Angiology. 2009 Feb-Mar;60(1):36-41. doi: 10.1177/0003319708317337. Epub 2008 May 27. PMID 18505746
- [Background] Gardner AW, Killewich LA, Montgomery PS, Katzel LI. Response to exercise rehabilitation in smoking and nonsmoking patients with intermittent claudication. J Vasc Surg. 2004 Mar;39(3):531-8. doi: 10.1016/j.jvs.2003.08.037. PMID 14981444
- [Background] Figueroa A, Park SY, Seo DY, Sanchez-Gonzalez MA, Baek YH. Combined resistance and endurance exercise training improves arterial stiffness, blood pressure, and muscle strength in postmenopausal women. Menopause. 2011 Sep;18(9):980-4. doi: 10.1097/gme.0b013e3182135442. PMID 21540753
- [Background] Brewer LC, Chai HS, Bailey KR, Kullo IJ. Measures of arterial stiffness and wave reflection are associated with walking distance in patients with peripheral arterial disease. Atherosclerosis. 2007 Apr;191(2):384-90. doi: 10.1016/j.atherosclerosis.2006.03.038. Epub 2006 May 26. PMID 16730015